CLINICAL TRIAL: NCT05437978
Title: "Sport on Prescription" in Primary Care for Patients With Long-term Illnesses: From General Practitioners' Prescriptions to the "Maison Sport Santé" System for Adapted Physical Activity
Brief Title: "Sport on Prescription" in Primary Care for Patients With Long-term Illnesses
Acronym: PRIMAPA-VAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too many missing data for primary outcome linked to patients stopping the program before the required visit
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-CHITS-001; 2022-A00712-41 (Other: ID-RCB)
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Chronic Illness
Keywords: Chronic disease; Adapted Physical Activity; Prescription; Quality of life
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted Physical Activity (APA) program called "Cap Sport Santé 83" (Experimental)
  Interventions: Other: "Cap Sport Santé 83" program

INTERVENTIONS:
Other: "Cap Sport Santé 83" program — In Var department (France), the " Maison Sport-Santé 83 " has set up a program called "Cap Sport Santé 83" to support patients who received a prescription to practice APA regularly. This program helps long-term illnesses patients to restart physical activity by considering their pathology. The "Cap Sport Santé 83" program is composed of 5 stages which aim to encourage adherence to APA practice by relying on the medical prescription system. Throughout the process, the patient is supervised and supported by the program's coordinator.

SUMMARY:
Adapted Physical Activity (APA) helps to prevent chronic diseases identified as major causes of mortality, particularly cardiovascular diseases and some cancers, according to the World Health Organization (WHO). However, in general population, physical activity levels are below recommendations for nearly 40% of french adults. In France, general practitioners are now authorised and encouraged to prescribe APA to long-term illness patients.

In Var department in France, the " Maison Sport-Santé 83 " has set up a program called "Cap Sport Santé 83" to support patients who received a prescription to practice APA on a regular basis. This program helps long-term illness patients to restart physical activity by considering their pathology.

The aim of this study is to evaluate " Maison Sport-Santé 83 " APA program effectiveness using a rigorous scientific methodology.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a long-term illness of any type, or a chronic illness, or risk factors (such as hypertension or obesity), or persons with decreasing independance and a stabilised clinical condition
* Aged 18 years old or over
* Able to express his/her consent prior to participation in the study
* Understanding french language
* Affiliated to or beneficiary of a social security regimen

Exclusion Criteria:

* Patient with a contraindication to physical activity
* Pregnant women
* Patient under judicial protection (guardianship, curatorship...) or safeguard of justice
* Any other reason that, in the opinion of the investigator, might interfere with the evaluation of the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the program impact on quality of life by the physical component of SF-36 questionnaire | 6 months
  A high score corresponds to better health/quality of life.

SECONDARY OUTCOMES:
To evaluate the program impact on quality of life by the mental health and physical components of SF-36 questionnaire | Up to 12 months
  A high score corresponds to better health/quality of life.
To evaluate physical activity by 6-minute walk test | Up to 12 months
  The 6-minute walk test allows to classify patients according to their functional capacity degree (4 categories: no limitation, minimal limitation, moderate limitation, severe limitation) by measuring the distance covered by patients in 6 minutes.
To evaluate physical activity by 30-Second Sit to Stand Test | Up to 12 months
  Patients will be asked to sit down and stand up without using arms, as many times as possible in 30 seconds. Number of completed repetitions will be recorded.
  The more repetitions the patient does, the greater the muscle power of the lower limbs.
Physical activity and sedentary behaviour measured by the Global Physical Activity Questionnaire (GPAQ) | Up to 12 months
  The GPAQ is an instrument to evaluate duration of vigorous and moderate physical activities covering 3 domains: activities at work, recreational domains and transport domains. Activity is calculated in MET value and classify patients according to 3 levels of physical activity defined as highly active, moderate and low.
Body composition measured by ultrasound and waist measurement. | Up to 12 months
  Total mass, percentage of fat mass, percentage of lean mass will be measured by ultrasound and recorded as well as waist measurement.
Heart rate and heart rate variability measured with a heart rate monitor | Up to 12 months
  Heart rate will be recorded
Quality of motivation to physical activity measured by the Motivation to Engage in Physical Activity in the Health Context Scale (EMAPS) | Up to 12 months
  The EMAPS is a motivation scale toward health-oriented physical activity in French which includes 6 components of motivation underlined by self-determination theory. The higher the component scores, the higher the form of motivation associated with that component.
To measure Body Mass Index (BMI) | Up to 12 months
  Weight and height will be recorded.
To measure Blood pressure by tensiometer | Up to 12 months
  Blood pressure will be recorded.
Physical activity and sedentary behaviour measured by accelerometry | Up to 6 months
  Accelerometry evaluate a subject's physical activity using sensors (accelerometers) that measure the body's accelerations and decelerations
Balance function | Up to 12 months
  Patient's balance will be assessed thanks to an equilibrium test on one foot. Time before equilibrium loss will be measured by means of a chronometer.
Hand muscle strength | Up to 12 months
  Hand muscle strength will be evaluated thank to a dynamometer which will have to be clutched as much as possible by the patient.
Trunk flexibility | Up to 12 months
  Trunk flexibility will be assessed through a forward bend test. Once the patient has reached his maximal position, the distance between ground and his fingertips will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie LAMOULERE, MD, Study Director — Maison Sport Santé 83
Locations (1):
- Maison Sport Santé 83, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No